CLINICAL TRIAL: NCT03377933
Title: The Effects of Compound Lactobacillus Acidophilus Has on Gastromicroecology and Combined With Tetracycline- and Furazolidone- Containing Quadruple Regimen as Rescue Treatment for Helicobacter Pylori Infection
Brief Title: The Effects Probiotic Has on Gastromicroecology and Combined With Quadruple Regimen for H Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yiqi Du (Other)
Responsible Party: Sponsor-Investigator, Yiqi Du, Vice Director of Department of Gastroenterology, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: chbs230023-1
Record Dates: First submitted 2017-12-01; First posted 2017-12-19 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Efficacy; Gastric Microbiota; Safety
Keywords: Helicobacter pylori; Probiotics; Efficacy; Safety; gastromicroecology

STUDY DESIGN:
Intervention Model Description: Single-center exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- probiotics and quadruple therapy (Experimental): Patients are given two-week compound Lactobacillus acidophilus probiotic (1 g t.i.d.), followed by a quadruple antibiotic regimen (esomeprazole [20 mg b.i.d.] + bismuth potassium citrate [220 mg b.i.d.] + tetracycline [750 mg b.i.d.] + furazolidone [100 mg b.i.d.]) for 10 days as rescue therapy.Meanwhile perform endoscopy and take gastric mucosa specimens for gene sequencing before and after the application of probiotic.
  Interventions: Other: Compound Lactobacillus acidophilus

INTERVENTIONS:
Other: Compound Lactobacillus acidophilus — Compound Lactobacillus acidophilus Tablet
  Other Names: Yi Jun Kang

SUMMARY:
This study assesses the efficacy and safety of treatment with two-week probiotics followed by a 10-day tetracycline- and furazolidone-containing quadruple regimen as rescue treatment for H. pylori infection. Eradication was evaluated using the 13C-urea breath test at 4 weeks after the end of therapy, and side effects were recorded. Besides study gene-level changes in the gastric microbiota following use of probiotics.

DETAILED DESCRIPTION:
Currently the infection rate of H. pylori is high. H. pylori infection has a close relationship with human diseases , Among the patients with H. pylori infection, 100% have active gastritis, <10% show H. pylori related dyspepsia, 15%~20% develop into peptic ulcer, <1% ultimately evolve into gastric malignant tumor. H. pylori gastritis has been defined as an infective disease. Eradication of H. pylori plays an important role in the cure, reversal and delay of these diseases.

With the widespread eradication of H. pylori, antibiotics resistance rates are increasing seriously. The resistance of antibiotics results in the increase of H. pylori eradication failure rate. Choosing a safe and effective scheme for patients who have failed multiple times is a challenge for the clinicians.

Besides, both domestic and international consensuses point that the application of some probiotics can reduce adverse effects through regulating gastric microenvironment, and it is still controversial about whether probiotics can inhibit H. pylori to increase the eradication rate.

Investigators previously retrospectively analyzed 30 patients with H. pylori eradication failures at least two times given two-week compound Lactobacillus acidophilus followed with 10-day tetracycline- and furazolone- containing quadruple regimen, the ITT eradication rate was 92.1%, and 94.6% PP analysis. Side effects were mild mainly including dizziness, dry mouth and skin rash occurred in eight patients.

ELIGIBILITY:
Inclusion Criteria:

* All included patients were 18 to 70 years-old; negative for the urea breath test at least 4 weeks after last eradication treatment; and experienced at least 2 H. pylori eradication failures.

Exclusion Criteria:

* Patients were excluded if they presented with a severe comorbidity or a malignant tumor; had a known history of allergy to the drugs in the therapeutic regimen; used nonsteroidal anti-inflammatory drugs (NSAIDs), antibiotic therapy, or bismuth salts up to 4 weeks before study inclusion; or were pregnant or breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
gene-level changes in the gastric microbiota | 2 weeks
  study gene-level changes through gene sequencing in the gastric microbiota following use of probiotics

SECONDARY OUTCOMES:
eradication rate of the therapy | 4 weeks
  using the 13C-urea breath test at 4 weeks after the end of therapy
the incidence of the adverse effects | 2 weeks, 4 weeks
  record the side effects on the 2 week, 4 week.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Qi Du, professor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
study protocal